CLINICAL TRIAL: NCT01719081
Title: Ultrasound for Sacroiliac Joint Injection: Evaluation of the Efficacy of Two Image-Guided Techniques for Sacroiliac Joint Injection
Brief Title: Sacroiliac Joint Injection: Comparison of Xray Versus Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-0880-AE
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Sacroiliac Joint Arthritis Causing Low Back Pain
Keywords: Sacroiliac Joint; Ultrasound; Fluoroscopy; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound Guided SIJ Injection (Experimental): Needle placement will be performed under US guidance. Fluoroscopy will be used to confirm needle placement prior to medication injection.
  Interventions: Procedure: Sacroiliac Joint Injection
- Xray Guided SIJ Injection (Active Comparator): Needle placement will be performed under fluoroscopy.
  Interventions: Procedure: Sacroiliac Joint Injection

INTERVENTIONS:
Procedure: Sacroiliac Joint Injection — Medication injected into the sacroiliac joint: Bupivicaine 3ml 0.25% with epinephrine 1/200,000 and Depo-Medrol 40mg.

SUMMARY:
This project involves the assessment of the efficacy of two different image guided techniques in patients with low back pain due to arthritis of the sacroiliac joint (SIJ). Intra-articular injection of local anesthetics and steroids is performed to relieve pain originating from the SIJ. Fluoroscopy has been used traditionally for image guidance for this procedure but there is a growing interest in use of ultrasound (US) for this procedure. US avoids radiation exposure to the patient and the health care team (HCT) and is less expensive. We aim to compare procedural efficacy related outcomes for SIJ injections performed using these image-guided modalities.

DETAILED DESCRIPTION:
The study is a prospective, randomized trial. Patients with low back pain which is diagnosed secondary to SIJ disease will be identified beforehand in clinic and offered a therapeutic joint injection. Informed consent will be obtained. Patients will be randomized for SIJ block with 3 mL of 0.25% bupivacaine with 1:200,000 epinephrine and 40 mg depomedrol using guidance with ultrasound or fluoroscopy. In both groups, confirmation of needle placement will be obtained using contrast injection imaging before the injection is performed. Record will be made of the number of times the needle is correctly placed into the articular space, as well as the number of attempts to do so. The final position of the needle will be recorded. Pain scores will be assessed before the procedure, as well as post-procedure at 24 and 72 hours, as well as 1 week, 1 month, and 3 months. Patients will keep a pain diary and will be followed up at 3 months time in clinic.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of SIJ disease on history: pain below the lumbo-sacral junction; pain with full weight-bearing on one leg; pain worse going down hills or inclines; very low back pain associated with groin pain and absence of lumbar symptoms
* Two positive responses to the following maneuver: FABER (flexion abduction and external rotation of hip), POSH (posterior shear test), REAB (resisted abduction)
* Baseline NRS pain score > or = to 4
* Refractory to oral analgesic therapy

Exclusion Criteria:

* ongoing litigation issues related to the patient's pain
* pregnancy
* allergy to steroids or local anesthetics
* multiple comorbidities
* BMI > 35

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Incidence of needle placement into SIJ | Assessed at time of injection
Pain - Numeric Rating Scale Score at 1 month | One month from time of injection

SECONDARY OUTCOMES:
Improvement of functional ability at 1 month | 1 month from time of injection
  Oswestry Disability Index completed at 1 month to determine level of disability
Patient Satisfaction | 1 month from time of injection
Average daily consumption of opioids at 1 month | 1 month from injection
Patient discomfort with procedure | Measured at time of procedure
Number of needle readjustments | Measured at time of procedure

OTHER OUTCOMES:
Assessment of complications | Until 3 months after procedure
  Complications assessed at any point until 3 months after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Anuj Bhatia, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada